CLINICAL TRIAL: NCT06667778
Title: Effectiveness of Osseodensification in Enhancing Implant Stability and Ridge Expansion in Esthetic Region (a Randomized Controlled Clinical Trial)
Brief Title: Osseodensification in Enhancing Implant Stability and Ridge Expansion in Esthetic Region
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant Lecturer of Dental Public Health and biostatistical consultanat, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0105-12
Record Dates: First submitted 2024-10-30; First posted 2024-10-31 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Dental Implant; Bone Expantion

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental)
  Interventions: Device: Osseodesification densah burs
- Control group (Active Comparator)
  Interventions: Device: Microdent

INTERVENTIONS:
Device: Osseodesification densah burs — Drill no. VT1525 (2mm) of densah burs will be used first in counter clockwise (in the osteotomy site).
  Then drill no. VT2535 (3mm) of densah burs will be used in counter clockwise to put 3.5mm implant diameter.
  Arms: Study group
Device: Microdent — No. 1 Microdent expander will be placed and screwed slowely (to avoid heat generation) into the osteotomy site till reaching the full desired length.
  N0. 2 microdent expander will be placed and screwed into the osteotomy site as the same step.
  Then no. 3 Microdent expander will be inserted for placing 3.5mm implant diameter
  Other Names: Conventional manual bone expanders
  Arms: Control group

SUMMARY:
Dental implants supported restorations have been widely accepted as one of the treatment modalities to replace missing teeth and to restore human masticatory function. Successful osseointegration from the clinical standpoint is a measured by implant stability, which occurs after implant integration. Osseodensification is a bio-mechanical site preparation technique. It utilizes a multi-fluted densifying bur technology that creates and expands a pilot hole without excavating significant amounts of bone tissue through a unique, highly controllable, fast, and efficient procedure with minimal heat elevation.

Aim of the study: Is to evaluate and compare the efficacy of using osseodensification compared to conventional bone expansion in implant stability and ridge expansion.

ELIGIBILITY:
Inclusion Criteria:

* Missing maxillary anterior tooth, having moderate horizontal ridge defect in which the alveolar ridge width is( 3-4) mm, and its height is not less than 10 mm.
* Presence of adequate keratinized mucosa.
* Patients with good oral hygiene.
* Patients are free from any systemic diseases that might affect healing.
* Presence of adequate inter-occlusal and mesiodistal space that permits placement of fixed prosthesis.

Exclusion Criteria:

* Heavy smokers and bad oral hygiene patients.
* Medically compromised patients that affecting placement of implant.
* Alcohol or drug abuse.
* Pregnant women.
* Patients suffering from osteoporosis.
* Current chemotherapy or radiotherapy.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2021-01-12 (Actual); Primary Completion 2021-09-28 (Actual); Study Completion 2021-09-28 (Actual)

PRIMARY OUTCOMES:
Change in implant stability | Baseline and 16 weeks
  Implant stability will be measured using the Ostell device.

SECONDARY OUTCOMES:
Change in bone density | Baseline and 16 weeks
  The patients will be examined radiographically using CBCT
Change in ridge expansion | Baseline and 16 weeks
  The patients will be examined radiographically using CBCT
Change in bone loss | Baseline and 16 weeks
  The patients will be examined radiographically using CBCT

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient Clinic of Periodontology and Oral medicine Department, Faculty of Dentistry, Alexandria University, Egypt, Alexandria, Egypt

REFERENCES:
- [Derived] Hammouda MA, Lotfy ME, Anwar SK. Effectiveness of osseodensification in enhancing implant stability and ridge expansion in esthetic zone: a randomized controlled clinical trial. Odontology. 2026 Jan 6. doi: 10.1007/s10266-025-01284-1. Online ahead of print. PMID 41493727